CLINICAL TRIAL: NCT06165614
Title: Self-administered Artesunate Pessaries for Treatment of Cervical Precancer in Kenya
Brief Title: Artesunate Pessaries (Vaginal Inserts) for Cervical Precancer in Kenya
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2236
Record Dates: First submitted 2023-11-21; First posted 2023-12-11 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Cervix Cancer; Cervix Neoplasm; Precancerous Conditions; Cervical Precancer
Keywords: vaginal pessaries; artesunate
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Uterine Cervical Dysplasia | interventions — Colposcopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Artesunate vaginal inserts/ pessaries (Experimental): Artesunate vaginal inserts/pessaries are used as a treatment for cervical precancerous lesions.
  Interventions: Drug: Artesunate pessary; Procedure: Colposcopy

INTERVENTIONS:
Drug: Artesunate pessary — Subjects will self-administer 200 mg of Artesunate pessary (vaginal insert) daily for 5 days, on weeks 1, 3, 5, 7.
Procedure: Colposcopy — Colposcopy is a procedure that allows close examination of the cervix, vagina, and vulva, performed on weeks 8 and 14.

SUMMARY:
To investigate the use of self-administered artesunate vaginal pessaries as treatment for cervical precancer in low and middle-income countries (LMIC). The central hypothesis of this study is that self-administered intravaginal Artesunate will be safe, and result in a clinical response among both HIV-positive and HIV-negative women with cervical precancer in LMICs.

DETAILED DESCRIPTION:
Despite being preventable, cancer of the cervix is a leading cause of cancer death in Kenya and other low- and middle-income countries (LMIC). Cervical cancer can be prevented if early changes in the cervix, called cervical precancer, are detected through screening, and adequately treated. Cervical precancer treatment includes a surgical procedure called Loop Electrosurgical Excision Procedure (LEEP), which removed the involved area of the cervix.

In countries like Kenya, this LEEP procedure is only available in referral hospitals which have trained consultants, and hence is difficult to access for most women who live in rural areas and away from tertiary facilities. Additionally, the LEEP procedure also increases the chance of a woman not being able to carry a pregnancy to full term, because the cervix is shorter after the procedure. For these reasons, alternative treatments, including self-administered treatments such as Artesunate are being investigated as alternative cervical precancer treatment that can be self-administered.

ELIGIBILITY:
Inclusion Criteria:

1. Cervical lesions referred for excision with CIN2/3 diagnosis on biopsy
2. Weight ≥50 kg
3. Agreement to use contraception (barriers or hormonal) through week 24 of the study if of childbearing age.
4. Ability and willingness to provide informed consent.

Exclusion Criteria:

1. Current pregnancy or breastfeeding status.
2. Current or past history of invasive cervical cancer.
3. History of total hysterectomy.
4. CD4 count less than 200 cells/mm3.
5. Presence of adenocarcinoma in situ on cervical biopsy
6. Currently receiving systemic chemotherapy or radiation therapy for another cancer
7. Current use of systemic immunosuppressants or steroids (>10 mg of prednisone or equivalent)
8. Have a medical comorbidity that in the opinion of the investigator would interfere with study participation.
9. Prior chemotherapy within 1 month prior to day 1 of study treatment
10. Male at birth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 17 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
the type, frequency, severity and duration of adverse events | From the first day of the study treatment to week 14 ( 8 weeks after artesunate use)
  Safety will be assessed by evaluating the type, frequency, severity, and duration of adverse events (AEs) using the U.S National Cancer Institute Common Terminology Criteria for Adverse Events, v5.0 (CTCAE 5.0).
  The NCI Common Terminology Criteria for Adverse Events is a descriptive terminology that can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.

SECONDARY OUTCOMES:
Adherence | From the first day of the study treatment to week 14 ( 8 weeks after artesunate use)
  Adherence will be evaluated based on participant self-report, returned packaging for used pessaries, and inspection of vaginal applicators under ultraviolet light for evidence of intravaginal insertion. A participant will be considered adherent if both methods support use of 80% (16 of 20) of the pessaries.
Change in lesion | From the first day of the study treatment to week 24
  Change in lesion size will be assessed by comparing colposcopic images of cervical lesions at baseline compared to the time of excision or week 24, whichever comes earlier, noting changes in the number and size of lesions and cervical quadrants involved. Blinded before and after treatment images will be evaluated by two gynecologists not involved in the study for evidence of a reduction in lesion size (Yes/No). A third gynecologist will be used as a tiebreaker if the two do not agree. The difference in proportions with the reduction in lesion size between the HIV-positive and HIV-negative groups will be reported.
Histologic regression | From the first day of the study treatment to week 24
  Histologic regression will be evaluated by comparing the initial diagnostic biopsy at study entry with the exit biopsy or excisional specimen final diagnosis. Participants who have complete regression at follow-up will have a confirmatory biopsy at the lesion site which will be used for final diagnosis. Regression will be defined as CIN1 or less in the resection or biopsy specimen. All specimens will be reviewed by a pathologist in-country and slides scanned for review by a 2nd pathologist at UNC. A 3rd pathologist will be utilized for consensus if the first two pathologists disagree. The difference in proportions with the histologic regression between the HIV-positive and HIV-negative groups will be reported.
Acceptability | At week 8
  Acceptability will be assessed using a questionnaire with study participants using Artesunate. Responses to questions will be graded on a Likert scale. The Likert scale has questions from 1 to 6. Higher scores represent better QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Chemtai Mungo, MD, MPH, FACOG, Principal Investigator — Lineberger Comprehensive Cancer Center, The University of North Carolina Chapel Hill
Locations (1):
- Lumumba Sub-County Hospital, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No
This can be requested and provided under reasonable request.

REFERENCES:
- [Derived] Guliam A, Sadana A, Opiyo E, Adundo F, Sorgi K, Agha E, Mungo C. Trying to Heal Without "Bringing Problems": Navigating Cervical Precancer Stigma in a Phase I Clinical Trial in Western Kenya. medRxiv [Preprint]. 2025 Dec 17:2025.10.24.25338728. doi: 10.1101/2025.10.24.25338728. PMID 41415498
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials